CLINICAL TRIAL: NCT03705091
Title: Non Contrast Magnetic Resonance Imaging to Measure Renal Transplant Perfusion and Fibrosis - Association With Function and Prognosis
Brief Title: MRI in Renal Transplantation
Acronym: TransRASL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN15RE038
Record Dates: First submitted 2018-03-03; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-02

CONDITIONS: End Stage Renal Disease; Renal Transplant Rejection; Kidney Transplant Failure and Rejection; Chronic Kidney Diseases
Keywords: Magnetic resonance imaging; Biomarkers; Arterial spin labelling; Diffusion weighted imaging; Renal transplantation
MeSH Terms: conditions — Kidney Failure, Chronic; Rejection, Psychology; Renal Insufficiency, Chronic | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transplant: Incident patients receiving a kidney transplant for end stage kidney disease. Patients will undergo functional magnetic resonance imaging at 2 months, 6 months and 12 months following transplantation.
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — ASL and DWI MRI

SUMMARY:
Renal transplantation is the optimal method of treatment for end stage kidney disease however median lifespan of a kidney transplant is around 15 years. Existing methods of measuring transplant function and structure from blood and urine markers are imperfect; renal biopsy is often performed but is invasive. Novel methods of investigating transplant function are therefore required and emerging renal MRI sequences including ASL and diffusion weighted imaging may yield helpful biomarkers. Investigators will recruit 20 patients in the first year after transplant and measure MRI biomarkers at three time points, with correlation to existing methods of measuring transplant function.

DETAILED DESCRIPTION:
Kidney transplantation remains the optimal therapy for patients with end stage kidney disease and is associated with significant improvements in life expectancy and quality of life compared to subjects receiving dialysis. Despite significant advances in our understanding of the immune system and development of drugs to prolong transplant function, a large number (Scottish Renal Registry data suggest between 23-35%) of transplants fail in the 10 years from operation. This may be due to a number of factors but is often due to development of transplant rejection, where the recipient's immune system damages the transplant. Early recognition and implementation of therapy is needed to dampen this response, reduce irreversible damage and preserve transplant function.

At present, transplant function and damage is measured using blood and urine tests. These are far from perfect markers because there is a delay between transplant damage and abnormalities of these tests. This time is vital for the short and long term survival of the transplant.

In the University of Glasgow, investigators have developed a new type of magnetic resonance imaging (MRI) which allows assessment of kidney blood flow and fibrosis (scarring) without the need for administration of harmful contrast agents. Arterial spin labelling magnetic resonance imaging (ASL MRI) is a non-invasive method of measuring renal perfusion using magnetised blood as endogenous contrast and investigators have validated this technique previously in both individuals with and without kidney disease. Diffusion tensor imaging (DTI) is another modality of non-contrast MRI which allows measurement of 'stiffness' of renal transplants, which represents long term scarring and fibrosis.

The investigators intend to follow up people receiving a kidney transplant for one year, collecting samples of blood, urine, and performing MR imaging at 3 time points, in order to investigate novel biomarkers of transplant function and dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Recent or pending kidney transplantation
* Written informed consent

Exclusion Criteria:

* Severe chronic liver, heart or lung disease
* Chronic infection
* Unable to give valid informed consent
* Known pregnancy or intent to conceive during the study period
* Any contraindicating to MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have either recently received, or are undergoing assessment for kidney transplantation, will be recruited. Those receiving live donor transplants undergo surgery electively and can be approached prior to the time of transplant. Those receiving kidney transplants from the waiting list represent the majority of transplant patients, and undergo surgery at unpredictable time points depending on the availability of organs. These individuals will be approached shortly after transplantation. They will be identified from the electronic medical record and approached at the transplant assessment clinic or on the transplant ward. A participant information sheet will be given and the patient contacted after one week to confirm or refute participation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-02-20 (Estimated); Study Completion 2019-03-20 (Estimated)

PRIMARY OUTCOMES:
Change in arterial spin labelling (ASL) | Measured at 2, 6, 12 months after transplant
  Renal perfusion measured by ASL MRI

SECONDARY OUTCOMES:
Change in apparent diffusion coefficient (ADC) | Measured at 2, 6, 12 months after transplant
  Renal fibrosis measured by diffusion weighted imaging (DWI) MRI

CONTACTS AND LOCATIONS:
Locations (1):
- University of Glasgow, Glasgow, Renfrewshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized participant data may be shared with collaborators in renal imaging after study completion. Images will not be shared.